CLINICAL TRIAL: NCT02013193
Title: Prospective, Randomized, Multicentre Clinical Study of the Hemoteq Ranger™ Paclitaxel-Coated PTA Balloon Catheter (Ranger DCB) in Comparison to Uncoated PTA Balloons in Femoropopliteal Lesions
Brief Title: Comparison of the Ranger™ Paclitaxel-Coated PTA Balloon Catheter and Uncoated PTA Balloons in Femoropopliteal Arteries
Acronym: RANGER-SFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemoteq AG (Industry)
Collaborators: CERES GmbH (Industry); coreLab Black Forest GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HTQ001-RangerSFA; CIV-13-07-011514 (Other: EUDAMED)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Artery Disease; Claudication; Atherosclerosis; Arteriosclerosis
Keywords: drug-coated balloon; drug-eluting balloon; peripheral artery disease; claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Atherosclerosis; Arteriosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranger(TM) Paclitaxel-coated balloon (Experimental): Index lesion treated with Ranger(TM) Paclitaxel-coated PTA balloon catheter (Ranger DCB)
  Interventions: Device: Ranger DCB
- uncoated PTA balloon (Active Comparator): Index lesion treated with an uncoated standard PTA dilatation balloon catheter selected upon investigator´s discretion
  Interventions: Device: uncoated PTA balloon

INTERVENTIONS:
Device: Ranger DCB — After successful pre-dilatation the index lesion is treated with one or two Ranger DCB devices that completely cover the lesion. If two devices are deployed, overlap shall be minimal.
  Arms: Ranger(TM) Paclitaxel-coated balloon
Device: uncoated PTA balloon — The index lesion is treated with one or more uncoated standard PTA balloons that completely cover the lesion.
  Arms: uncoated PTA balloon

SUMMARY:
The primary objective of this study is to prove the superior performance of the Ranger™ paclitaxel-coated PTA balloon catheter for angioplasty for femoropopliteal artery lesions when compared to non-coated balloons at six months post-procedure when comparing Late Lumen Loss (LLL). Study statistical hypothesis: The %-mean loss of luminal diameter as assessed by angiography at six months follow-up after treatment of the femoropopliteal artery with Ranger DCB study devices is lower than the %-mean loss of luminal diameter after treatment with uncoated PTA balloon control devices.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 18 or older
* Subject is willing and able to provide informed consent
* Subject is available to attend all required follow-up visits
* Subject has a clinically significant symptomatic leg ischemia requiring treatment
* Subject has a Rutherford clinical category of 2-4
* If the index lesion is restenotic, the prior PTA must have been >30 days prior to treatment in the current study
* Only one lesion per limb can be treated under this protocol.
* Successful intraluminal wire crossing of the target lesion
* Index lesion is a clinically and hemodynamically significant stenotic or restenotic lesion located in the native nonstented superficial femoral artery or proximal popliteal artery
* Degree of stenosis 70% or more, by visual assessment
* Lesion length between 20 mm and 150 mm
* At least one patent infrapopliteal artery to the foot of the index limb

Exclusion Criteria:

* Subjects who have undergone prior vascular surgery of the femoropopliteal artery in the index limb to treat atherosclerotic disease
* History of major amputation in the same limb as the target lesion
* Presence of aneurysm in the target vessel
* Acute ischemia and/or acute thrombosis in any artery of the lower limbs
* Acute Myocardial Infarction within 30 days before the index procedure
* Persistent, intraluminal thrombus of the proposed target lesion post-thrombolytic therapy
* Known hypersensitivity or contraindication to contrast dye that cannot be adequately pre-medicated
* Known allergies against Paclitaxel or other components of the used medical devices
* Intolerance to antiplatelet, anticoagulant, or thrombolytic medications that would be administered during the trial
* Platelet count <100,000 mm3 or >600,000 mm3
* Concomitant renal failure with a serum creatinine >2.0 mg/dL
* Receiving dialysis or immunosuppressant therapy
* Life expectancy of less than one year
* Women of child-bearing potential must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.
* Woman who is pregnant or nursing.
* Previously planned stenting of the index lesion
* Use of adjunctive therapies (debulking, laser, cryoplasty, re-entry devices)
* Planned or expected procedures (cardiac, aorta, peripheral) within 30 days after the index procedure
* Presence of outflow lesions requiring intervention within 30 days of the index procedure
* Perforated vessel as evidenced by extravasation of contrast media
* Heavily calcified target lesions resistant to PTA
* Current participation in another drug or device trial that has not completed the primary endpoint, that may potentially confound the results of this trial, or that would limit the subject's compliance with the follow-up requirements
* Current participation in any study using drug-coated/drug-eluting technologies
* Current participation in any study using drug-coated/drug-eluting technologies
* Target lesion with in-stent restenosis (any stent or stent-graft)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
in-segment late lumen loss | six months
  In-segment late lumen loss (LLL) of the treated segment after PTA using the Ranger™ paclitaxel-coated PTA balloon, in comparison to the LLL after PTA using an uncoated balloon, as observed by angiography at six months post-index procedure.

SECONDARY OUTCOMES:
technical success | during index procedure, less 1 hour
  The ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%.
procedural success | within 24 hours of index procedure
  Technical success with no MAE noted within 24 hours of the index procedure.
primary patency | six months
  Percentage of lesions that reach endpoint without a hemodynamically significant stenosis on duplex ultrasound (DUS) and without target lesion revascularization (TLR) or bypass of the target lesion to maintain or restore patency.
primary patency | twelve months
  Percentage of lesions that reach endpoint without a hemodynamically significant stenosis on DUS and without TLR or bypass of the target lesion to maintain or restore patency.
assisted primary patency | six months
  Percentage of lesions without TLR and those with TLR (not due to complete occlusion or bypass) that reach endpoint without restenosis.
assisted primary patency | twelve months
  Percentage of lesions without TLR and those with TLR (not due to complete occlusion or bypass) that reach endpoint without restenosis.
secondary patency | six months
  Percentage of lesions with TLR for occlusion that reach endpoint without restenosis.
secondary patency | twelve months
  Percentage of lesions with TLR for occlusion that reach endpoint without restenosis.
binary restenosis rate | six months
  Binary restenosis defined as > 50% diameter stenosis via peak systolic velocity ratio (PSVR) > 2.4 via duplex ultrasound and assessed by the core lab.
binary restenosis rate | twelve months
  Binary restenosis defined as > 50% diameter stenosis via peak systolic velocity ratio (PSVR) > 2.4 via duplex ultrasound and assessed by the core lab.
clinical success | pre-discharge, estim. 1-2 days post-index procedure
  Positive change (by +1 or more) of Rutherford category at pre-discharge post-index-procedure as compared to baseline.
clinical success | six months
  Positive change (by +1 or more) of Rutherford category at six months (plus or minus 30 days) post-index-procedure as compared to baseline.
clinical success | twelve months
  Positive change (by +1 or more) of Rutherford category at twelve months (plus or minus 30 days) post-index-procedure as compared to baseline.
hemodynamic success | pre-discharge, estim. 1-2 days post-index procedure
  positive change in Ankle-Brachial Index (ABI) at pre-discharge as compared to baseline
hemodynamic success | six months
  positive change in ABI at six months (plus or minus 30 days) as compared to baseline
hemodynamic success | twelve months
  positive change in ABI at twelve months (plus or minus 30 days) as compared to baseline
change in quality of life | six months
  Change in functional status measured by changes in the Walking Impairment Questionnaire (WiQ) and general health-related quality of life measured by changes in SF-12 and EQ5D scores at six months (plus or minus 30 days) as compared to baseline.
change in quality of life | twelve months
  Change in functional status measured by changes in the Walking Impairment Questionnaire (WiQ) and general health-related quality of life measured by changes in SF-12 and EQ5D scores at twelve months (plus or minus 30 days) as compared to baseline.
change in quality of life | 24 months
  Change in general health-related quality of life measured by changes in SF-12 and EQ5D scores at 24 months (plus or minus 30 days) as compared to baseline.
change in quality of life | 36 months
  Change in general health-related quality of life measured by changes in SF-12 and EQ5D scores at 36 months (plus or minus 30 days) as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, M.D., Principal Investigator — University Leipzig
Locations (11):
- Medical University, AKH, Vienna, Austria
- France (3):
  - CHU Caen Côte de Nacre, Caen
  - Hopital Europeen Georges-Pompidou (HEGP), Paris
  - Clinique Pasteur Toulouse, Toulouse
- Germany (7):
  - Klinikum Arnsberg, Arnsberg
  - Segeberger Kliniken, Bad Segeberg
  - Klinikum Darmstadt GmbH, Darmstadt
  - CardioVascular Center, Frankfurt
  - Universitätsklinikum Leipzig, Leipzig
  - Park-Krankenhaus, Leipzig
  - Universitätsklinikum, Marburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bausback Y, Willfort-Ehringer A, Sievert H, Geist V, Lichtenberg M, Del Giudice C, Sauguet A, Diaz-Cartelle J, Marx C, Strobel A, Schult I, Scheinert D; RANGER SFA Investigators. Six-Month Results From the Initial Randomized Study of the Ranger Paclitaxel-Coated Balloon in the Femoropopliteal Segment. J Endovasc Ther. 2017 Aug;24(4):459-467. doi: 10.1177/1526602817710770. Epub 2017 May 31. PMID 28558502